CLINICAL TRIAL: NCT04223583
Title: Study on the Treatment of Soft Tissue Sarcoma With First-line Chemotherapy Failure by Anrotenil Hydrochloride Capsule
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, YaoWeitao, Chief physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019212
Record Dates: First submitted 2019-09-26; First posted 2020-01-10 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Soft Tissue Sarcomas
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anrotenil hydrochloride capsule (Experimental): Anrotenil hydrochloride capsule was used to treat soft tissue sarcomas with first-line chemotherapy failure (doxorubicin + ifosfamide). Oral administration was conducted on an empty stomach before breakfast (12mg), and the drug was discontinued for 2 weeks for one week (3 weeks for one cycle) until the disease progressed or became intolerable.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — The standard first-line chemotherapy regimen (adriamycin + ifosfamide) failed
  Other Names: Oral administration of single drug on an empty stomach

SUMMARY:
Soft tissue sarcoma STS is a group of malignant tumors derived from connective tissue other than bone and cartilage. It can occur in any part of the body at any age, and there is no significant gender difference.According to pathological classification, STS has 19 tissue types and more than 50 disease subtypes.Currently, surgical resection, radiotherapy and drug therapy are the main treatment methods.But about 50% of the patients with distant metastasis happened not the surgical removal of, quite a number of in patients with distant metastasis after died of disease progression 8-12 months in drug treatment of soft tissue sarcoma, the current widely used chemotherapy regimens for ADM/IFO single-agent or joint IFO ADM is a line of chemotherapy, in addition, paclitaxel, gemcitabine, dorsey race, it was also used for soft tissue sarcomas of second-line chemotherapy scheme, however, for some special subtypes of sarcoma,Such as myxoid liposarcoma, pleomorphic rhabdomyosarcoma, leiomyosarcoma, glandular soft tissue sarcoma and superficial malignant fibrous histiocytoma, are not sensitive to chemotherapy or low sensitivity.Therefore, how to improve the survival rate of these patients is an urgent problem to be solved.

Anlootinib hydrochloride is a multi-target tyrosine kinase inhibitor that has shown good efficacy in solid tumors such as NSCLC, ovarian cancer, soft tissue tumors, and medullary thyroid cancer.Especially in the field of soft tissue sarcomas, the results of phase IIb clinical data were satisfactory.Therefore, Investigator plan to conduct the study of anrotenil hydrochloride capsule for the treatment of soft tissue sarcomas with first-line chemotherapy failure (anthracycline)

ELIGIBILITY:
Inclusion Criteria:

1. The patients volunteered to participate in this study and signed the informed consent;
2. Pathologically confirmed advanced soft tissue sarcomas with at least one measurable lesionMainly including Synovial sarcoma (Synovial sarcoma), Leiomyosarcoma (Leiomyosarcoma), gland Alveolar soft tissue sarcoma (Alveolar soft part sarcoma), Undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma (Undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma), liposarcoma (AdipocyticEpithelial sarcoma, Fibrosarcoma, Clear cell sarcoma, Epithelioid sarcoma, and other Tumors.Except for:Malignant peripheral nerve sheath tumor, Undifferentiated sarcoma, Rhabdomyosarcoma, chondrosarcoma, Osteosarcoma, dermato-fibrosarcomaProtuberans, gastrointestinal stromal tumor, Primitive neuroectodermal tumor, Inflammatory myofibroblastic tumor, Malignant mesothelioma.
3. Patients who have failed treatment with at least one or two line chemotherapy regimen (doxorubicin + ifosfamide, gemcitabine + docetaxel) within the last 6 months (except for acinar soft tissue sarcoma);[note: treatment failure refers to the occurrence of disease progression or intolerance during treatment or within 3 months of the last treatment]
4. 18 ~ 70 years old;ECOG PS score is 0~1;Expected survival beyond 3 months;
5. Patients who are effective with other targeted drugs, but have drug resistance and disease progression, and stop taking drugs for more than 4 weeks;
6. Major organ functions meet the following criteria within 7 days before treatment:

   1. blood routine examination standard (in the condition of no blood transfusion within 14 days) :

      * hemoglobin (HB) ≥90g/L;
      * absolute value of neutrophils (ANC)≥1.5×109/L;
      * platelet (PLT) ≥80×109/L
   2. biochemical examination shall meet the following standards:

      * total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (ULN);
      * alanine aminotransferase (ALT) and aspartate aminotransferase AST≤ 2.5×ULN, if accompanied by liver metastasis, ALT and AST≤5×ULN;
      * serum creatinine (Cr)≤1.5×ULN or creatinine clearance rate CCr≥60ml/min;
   3. doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).
7. Women of childbearing age should agree that they must obtain a certain amount during the study period and within 6 months after the study Use contraceptives (such as intrauterine devices, birth control pills or condoms);Negative serum or urine pregnancy test within 7 days before study enrollment and must be non-lactating;Men should agree to patients who must use contraception during the study period and within 6 months of the end of the study period.

Exclusion Criteria:

1. Patients who have previously used anlotinib hydrochloride capsules;
2. With pleural effusion or ascites, cause respiratory syndrome (≥CTC AE grade 2 dyspnea);
3. Patients who have received targeted therapy of vascular endothelial growth inhibitors, such as sunitinib, sorafenib, imatinib, bevacizumab, famitinib, apatinib, reagfenib and other drugs, have failed to respond to treatment.Other malignancies were present or present at the same time within 4.5 years, except cured carcinoma in situ of the cervix, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
4. Systemic antitumor therapy, including cytotoxic therapy, immunotherapy, or mitomycin C, was planned for the first 4 weeks of the group or in this study.Radiotherapy was performed in the first 4 weeks or in the second 2 weeks before the grouping.
5. Unrelieved toxic reactions above CTC AE(4.0) level 1 due to any previous treatment, excluding hair loss;
6. Having multiple factors affecting oral medications (such as inability to swallow, chronic diarrhea and intestinal obstruction);
7. Patients with brain metastasis with symptoms or symptom control time less than 2 months;
8. Patients with any serious and/or uncontrolled illness, including:

   1. Patients with unsatisfactory blood pressure control (systolic blood pressure ≥ 150 mmHg, diastolic blood pressure ≥ 100 mmHg);
   2. Patients with grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTc≥480ms) and grade ii or above congestive heart failure (New York heart association grade (NYHA));
   3. Active or uncontrolled severe infection (≥ grade CTC AE 2 infection);

      * Patients with cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis should receive antiviral treatment;
      * Renal failure requires hemodialysis or peritoneal dialysis;
9. Patients with any serious and/or uncontrolled illness, including:

   1. a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation;
   2. poor diabetes control (FBG > 10mmol/L);
   3. the urine routine indicated that urine protein ≥++, and confirmed the 24-hour urine protein quantitative > 1.0g.
   4. patients with seizures requiring treatment;
10. Significant surgical treatment, open biopsy or significant traumatic injury received within 28 days prior to grouping;
11. Any physical signs or history of bleeding, regardless of severity;Unhealed wounds, ulcers or fractures were found in patients with any bleeding or bleeding event ≥CTCAE level 3 within 4 weeks before grouping;
12. 6 months in the event of overactive/venous thrombosis, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism;
13. Having a history of abuse of psychotropic substances and being unable to quit or having mental disorders;
14. Participated in clinical trials of other anti-tumor drugs within four weeks; According to the researchers' judgment, there are concomitant diseases that seriously endanger patients' safety or prevent patients from completing the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Median progression-free survival（mPFS） | up to 12 months
  There are and only 50% of individuals who survive this time

SECONDARY OUTCOMES:
Objective response rate（ORR) | 2 years
  The percentage of patients whose tumors have shrunk to a certain amount of time and stayed that way for a certain amount of time

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, Deputy director, Study Chair — Henan Cancer Hospital
Locations (1):
- Affiliated Cancer Hospital of Zhengzhou University&Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
In order to better conduct clinical studies and ensure the prospective and timeliness of the studies, patients' IPD will be kept confidential.